CLINICAL TRIAL: NCT00701207
Title: Modulation of Pulmonary Sarcoidosis by Nicotinic Acetylcholine Receptors
Brief Title: Study of Nicotine Patches in Patients With Sarcoidosis
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Elliott Crouser MD (Other)
Collaborators: American Thoracic Society (Other)
Responsible Party: Sponsor-Investigator, Elliott Crouser MD, Medical Director, Intensive Care Unit, UHE, Ohio State University
Organization: Ohio State University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008H0006; S-07-006 (Other Grant/Funding Number: American Thoracic Society)
Record Dates: First submitted 2008-06-17; First posted 2008-06-19 (Estimated); Last update posted 2021-11-08 (Actual); Status verified 2021-11

CONDITIONS: Pulmonary Sarcoidosis
Keywords: To determine if nicotine treatment reduces lung inflammation
MeSH Terms: conditions — Sarcoidosis, Pulmonary | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 2. (No Intervention): control group-no intervention
- 3 (No Intervention): Healthy control group-blood and sputum samples
- 1. (Experimental): nicotine patch; transdermal patch 7mg, 14 mg., 21 mg. 3 months
  Interventions: Drug: nicotine patch

INTERVENTIONS:
Drug: nicotine patch — daily transdermal patch 7 mg, 14mg, 21 mg. 3 months
  Other Names: Habitrol QC
  Arms: 1.

SUMMARY:
The purpose of this study is to compare peoples with disease (sarcoidosis) to those without disease. We want to see if people with sarcoidosis have a different immune response to those people without disease.

The goal of this study is to see if the nicotine patch is an anti-inflammatory treatment for sarcoidosis.

DETAILED DESCRIPTION:
Until recently, there was no good explanation for the fact that smoking cigarettes actually reduces the risk of sarcoidosis. Research studies have shown that the nicotine, a common component of cigarette smoke, strongly suppresses the immune system and reduces the type of inflammation that is characteristic of sarcoidosis in the lungs. We propose that nicotine treatment, administered in the form of a skin patch, will reduce the severity of lung disease in patients with sarcoidosis. Sarcoidosis patients who volunteer to participate in this study will submit standardized questionnaires relating to their quality of life and the severity of their shortness of breath before and after treatment. We will also compare objective measures of lung function, radiographic parameters, and the severity of lung inflammation. We predict that nicotine treatment will reduce the severity of sarcoidosis symptoms, improve lung function, and resolve lung inflammation. If our hypothesis is proven to be correct in this relatively small group of patients, we will perform additional studies in a larger group of patients and will consider the features of sarcoidosis patients that predict a favorable response to nicotine and other nicotine-like drugs. If nicotine is ultimately found to be an effective treatment for sarcoidosis, it may replace some of the existing treatments which are frequently ineffective and have unacceptable side-effects.

ELIGIBILITY:
Inclusion Criteria:

* • Symptomatic (active) granulomatous lung disease (radiographic stage II or III disease) at least 6 months after the diagnosis. This selects patients that have the chronically active variant of sarcoidosis and will likely require long-term treatment (33).

Exclusion Criteria:

* • Active smokers,

  * Previous splenectomy,
  * Those requiring high-dose immunosuppression [i.e., ≥ 0.2 mg/kg/day prednisone (or equivalent) or > 10 mg/week methotrexate or requires second line cytolytic agents (e.g., cyclophosphamide, azathioprine) or anti-TNF treatments (e.g., thalidomide, anti-TNF antibodies, etc.)] to control disease activity.
  * We will also exclude patients at high risk of complications relating to the use of nicotine. This will include patients with a known intolerance of nicotine or those with active cardiac or central nervous system disease who are at higher risk of cardiac arrhythmias or seizures.
  * We will also exclude patients with extensive pulmonary fibrosis based upon lung biopsy or high resolution CT scan criterion

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2008-07; Primary Completion 2010-12-31 (Actual); Study Completion 2010-12-31 (Actual)

PRIMARY OUTCOMES:
To determine if nicotine treatment reduces lung inflammation. | 3 months
  Normalization of immune response

SECONDARY OUTCOMES:
To determine if expression of α7 nAChR on monocytes/macrophages derived from the blood/lungs correlates with the severity of pulmonary sarcoidosis. | 3 months
  Improvement in FVC

CONTACTS AND LOCATIONS:
Overall Officials: Elliott D. Crouser, M.D., Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

REFERENCES:
- [Background] Julian MW, Shao G, Schlesinger LS, Huang Q, Cosmar DG, Bhatt NY, Culver DA, Baughman RP, Wood KL, Crouser ED. Nicotine treatment improves Toll-like receptor 2 and Toll-like receptor 9 responsiveness in active pulmonary sarcoidosis. Chest. 2013 Feb 1;143(2):461-470. doi: 10.1378/chest.12-0383. PMID 22878868